CLINICAL TRIAL: NCT00806520
Title: Use of Continuous Glucose Monitoring Combined With Ambulatory Glucose Profiles to Characterize Glycemic Control Addendum to: A Randomized, Double-Blind, Parallel-Group, Multicenter Study to Compare the Glycemic Effects, Safety, and Tolerability of Exenatide Long-Acting Release to Those of Sitagliptin and Pioglitazone in Subjects With Type 2 Diabetes Mellitus Treated With Metformin (Study BCB106)
Brief Title: Use of Continuous Glucose Monitoring Combined With Ambulatory Glucose Profiles to Characterize Glycemic Control
Status: Completed | Type: Observational
Sponsor: HealthPartners Institute (Other)
Collaborators: Amylin Pharmaceuticals, LLC. (Industry)
Responsible Party: Sponsor
Other Study IDs: 03671-08-C
Record Dates: First submitted 2008-12-08; First posted 2008-12-10 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2011-08

CONDITIONS: Type 2 Diabetes
Keywords: Continuous Glucose Monitoring; Exenatide Once Weekly or; Januvia or; Actos
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Obtain Continuous Glucose Monitoring (CGM) data from individuals taking exenatide LAR, sitagliptin, or pioglitazone. The CGM measurements collected will help determine the characteristics of glucose control prior to treatment and during treatment.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* type 2 diabetes
* A1c 7.1 - 11
* BMI 25 - 45
* stable weight for 3 months before screening
* fasting glucose < 280 at screening
* stable dose of metformin for at least 2 months before screening
* not being treated with or on a stable dose of hormone replacement therapy, oral contraceptives, anti-hypertensive agents, lipid lowering agents, thyroid replacement therapy, anti-depressants, drugs known to affect body weight
* male or female, non-lactating, non-pregnant and willing to use birth control
* lab values that are not clinically significant at screening
* physical exam and ECG that are not clinically significant at screening
* able to read, understand, and sign consent form

Exclusion Criteria:

* liver disease
* renal disease
* cardiovascular disease
* gastroparesis
* cancer within 5 years of screening
* macular edema
* chronic infections
* drug or alcohol abuse
* fasting triglycerides > or = 600 at screening
* previous exposure to exenatide LAR
* has donated blood within 60 days of screening or is planning to donate during the study
* has had a major surgery or blood transfusion within 2 months before screening
* is currently being treated or is expecting to be treated with Byetta, Januvia, SU, TZD, GLP-1 analog, alpha-glucosidase inhibitor, meglitinide, nateglinide, symlin, insulin, systemic corticosteroids, lopid or rifampin
* has received an investigational drug within 1 month before screening
* has allergies or hypersensitivity to any component of the study drug
* has previously had an adverse event related to TZD or Januvia
* is an immediate family member of the study sight or directly affiliated
* is employed by Amylin, Lilly or Alkermes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants in the Amylin BCB106 Protocol Main Study
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2008-04; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard M. Bergenstal, MD, Principal Investigator — International Diabetes Center at Park Nicollet; Roger S. Mazze, PhD, Principal Investigator — International Diabetes Center at Park Nicollet; Robert M. Cuddihy, MD, Principal Investigator — International Diabetes Center at Park Nicollet; Elinor (Ellie) S. Strock, APRN, BS,CDE, Principal Investigator — International Diabetes Center at Park Nicollet
Locations (5):
- United States (5):
  - Joslin Diabetes Center, Boston, Massachusetts
  - International Diabetes Center, Minneapolis, Minnesota
  - Palm Medical Group, Las Vegas, Nevada
  - University of North Carolina Diabetes Care Center, Durham, North Carolina
  - Rockwood Clinic, Spokane, Washington